CLINICAL TRIAL: NCT00153088
Title: A Randomised, Double-blind, Placebo-controlled, Multicenter Trial to Investigate the Preventive Effect of BIBR277 (Telmisartan) in Diabetic Nephropathy on Transition From Incipient to Overt Nephropathy - Incipient to Overt : Angiotensin 2 Receptor Blocker, Telmisartan, Investigation on Type 2 Diabetic Nephropathy (INNOVATION Study -
Brief Title: INNOVATION Study - Telmisartan (Micardis) in Incipient Diabetic Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.413
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Telmisartan

INTERVENTIONS:
Drug: Telmisartan capsule 40 mg
Drug: Placebo
Drug: Telmisartan capsule 80 mg

SUMMARY:
The aim of this study is to compare the preventive effect of Telmisartan(Micardis) versus placebo control on the transition to overt nephropathy in patients with diabetic nephropathy manifesting microalbuminuria associated with type II diabetes, and to evaluate the efficacy and safety of Telmisart (Micardis, Gliosartan, Kinzal, Kinzalmono, Predxal, Pritor, Samertan, Telmisartan) for diabetic nephropathy patients.

DETAILED DESCRIPTION:
A prospective, randomised, double-blind, multicentric and comparative study to investigate, on a long-term basis, the preventive effect on the transition to overt nephropathy and the safety of Telmisartan (Micardis) against placebo in patients with diabetic nephropathy, manifesting microalbuminuria associated with type II diabetes.

Study Hypothesis:

The hypothesis is that Telmisartan (Micardis) at 40 mg or 80 mg versus placebo control in patients with concurrent type II diabetic mellitus or diabetic nephropathy demonstrating microalbuminuria, has the preventive effect on transition from incipient to overt nephropathy.

Comparison(s):

The primary endpoint is defined as the transition from incipient to overt nephropathy, and the non-transition curve will be demonstrated based on the Kaplan-Meier method. The evaluation criteria for the point to transition to overt nephropathy is defined as urinary albumin to creatinine ratios at consecutive 2 measuring points increasing over 300 mg/g-Creatinine and excess 30% increase comparing with the baseline value. The curve of non-transition will be compared with Logrank test. Those in BIBR277 groups are sequentially compared with that in the placebo group by the closed testing procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients who are able to visit the study site throughout the run-in period
2. Aged 30 and 74 years
3. Type II diabetes mellitus
4. Patients with urinary albumin to creatinine ratios within the following ranges at 2 measuring points during the run-in period 1) the first-morning voided urine, iin the range of 100 to 300 mg/g Creatinine 2) < 100 mg/g Creatinine at either point of Visit 2 or 3, but in the range of 100 to 300 mg/g Creatinine at follow-up
5. Serum creatinine level of < 1.5 mg/dL in male and < 1.3 mg/dL in female
6. Normotensive or hypertensive patients
7. Patients taking AT1 antagonists or ACE inhibitors at screening, but are able to stop those drugs during the study
8. Patients who are able to provide written informed consent in accordance with the Good Clinical Practice (GCP) and other relevant laws such as the Pharmaceutical Affairs Law

Exclusion Criteria:

1. Age of onset of type 2 diabetes is < 30 years
2. Type I diabetes
3. Urinary albumin to creatinine ratio of > 300 mg/g Creatinine
4. HbA1c 9%
5. Seated SBP 180 mmHg or DBP 110 mmHg
6. Findings suggesting a renal disease other than diabetic nephropathy; such as post renal transplantation, history of non-diabetic renal disease, marked haematuria, complication of urinary tract infection
7. Cardiovascular diseases:

   * Patients with unstable angina, myocardial infarction, CABG, PTCA within 6 months before
   * CHF with NYHA III-IV
   * TIA within 6 months
   * Stroke within 6 months
   * AV block (grade II-III) or AF
   * Serious arrhythmia
   * Known or suspected secondary HT
8. History of angioedema during administration of ARB/ACE-i
9. Hypersensitivity
10. History of sudden exacerbation of renal function due to ARB/ACE-i
11. Markedly poor bile secretion
12. Hepatic dysfunction: SGPT (ALT) or SGOT (AST) 100 IU/L
13. Serum potassium level < 3.5 mEq/L or 5.1 mEq/L
14. Unable to discontinue ARB/ACE-i
15. Require prolonged administration of any medications affecting blood pressure, except diuretics, or blockers, and CCB
16. Untreated sodium depletion
17. Pre-menopausal females who meet any one of the following:

    * Pregnant or possibly pregnant
    * Breast-feeding
    * Hope to be pregnant during the study period
    * Even when a patient is confirmed not to meet the above criteria at the start of the study, a female patient who has the potential to be pregnant during the study is to undergo pregnancy tests. If the result turns positive, the study medication should be discontinued.
18. Malignant tumour or other diseases requiring oral or injection immunosuppressants
19. Non-compliance
20. History of drug or alcohol abuse
21. Participated in other clinical studies within 3 months
22. Any other conditions investigators judged as ineligible

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2003-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11

PRIMARY OUTCOMES:
Non-transition to overt nephropathy

SECONDARY OUTCOMES:
Change in renal parameters Composite endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Nippon Boehringer Ingelheim Co., Ltd.
Locations (107):
- Japan (107):
  - Boehringer Ingelheim Investigational Site, Adachi-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Amagasaki, Hyogo
  - Boehringer Ingelheim Investigational Site, Arakawa-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Asaguchi-gun, Okayama
  - Boehringer Ingelheim Investigational Site, Asahi, Chiba
  - Boehringer Ingelheim Investigational Site, Asahikawa, Hokkaido
  - Boehringer Ingelheim Investigational Site, Asahikwa, Hokkaido
  - Boehringer Ingelheim Investigational Site, Atami, Shizuoka
  - Boehringer Ingelheim Investigational Site, Atsugi,Kanagawa
  - Boehringer Ingelheim Investigational Site, Chikugo, Fukuoka
  - Boehringer Ingelheim Investigational Site, Chisagata-gun, Nagano
  - Boehringer Ingelheim Investigational Site, Chitose, Hokkaido
  - Boehringer Ingelheim Investigational Site, Chiyoda, Tokyo
  - Boehringer Ingelheim Investigational Site, Chiyoda-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Ebina, Kanagawa
  - Boehringer Ingelheim Investigational Site, Fujisawa, Kanagawa
  - Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - Boehringer Ingelheim Investigational Site, Fukuyama, Hiroshima
  - Boehringer Ingelheim Investigational Site, Funabashi, Chiba
  - Boehringer Ingelheim Investigational Site, Furukawa, Miyagi
  - Boehringer Ingelheim Investigational Site, Gifu, Gifu
  - Boehringer Ingelheim Investigational Site, Gobo, Wakayama
  - Boehringer Ingelheim Investigational Site, Hachioji, Tokyo
  - Boehringer Ingelheim Investigational Site, Hakodate, Hokkaido
  - Boehringer Ingelheim Investigational Site, Hanamaki, Iwate
  - Boehringer Ingelheim Investigational Site, Hannan, Osaka
  - Boehringer Ingelheim Investigational Site, Hashima-gun, Gifu
  - Boehringer Ingelheim Investigational Site, Hatsukaichi, Hiroshima
  - Boehringer Ingelheim Investigational Site, Hirakata, Osaka
  - Boehringer Ingelheim Investigational Site, Hitachiota, Ibaragi
  - Boehringer Ingelheim Investigational Site, Ichinomiya, Aichi
  - Boehringer Ingelheim Investigational Site, Iida, Nagano
  - Boehringer Ingelheim Investigational Site, Ikeda, Osaka
  - Boehringer Ingelheim Investigational Site, Inashiki-gun, Ibaragi
  - Boehringer Ingelheim Investigational Site, Isehara, Kanagawa
  - Boehringer Ingelheim Investigational Site, Isezaki, Gunma
  - Boehringer Ingelheim Investigational Site, Itami, Hyogo
  - Boehringer Ingelheim Investigational Site, Izumisano, Osaka
  - Boehringer Ingelheim Investigational Site, Kamakura, Kanagawa
  - Boehringer Ingelheim Investigational Site, Kamogawa, Chiba
  - Boehringer Ingelheim Investigational Site, Katsushika-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Kawagoe, Saitama
  - Boehringer Ingelheim Investigational Site, Kawaguchi, Saitama
  - Boehringer Ingelheim Investigational Site, Kawasaki, Kanagawa
  - Boehringer Ingelheim Investigational Site, Kisarazu, Chiba
  - Boehringer Ingelheim Investigational Site, Kita-katushika-gun, Saitama
  - Boehringer Ingelheim Investigational Site, Kita-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Kitami, Hokkaido
  - Boehringer Ingelheim Investigational Site, Kobe, Hyogo
  - Boehringer Ingelheim Investigational Site, Kochi, Kochi
  - Boehringer Ingelheim Investigational Site, Kodaira, Tokyo
  - Boehringer Ingelheim Investigational Site, Komaki, Aichi
  - Boehringer Ingelheim Investigational Site, Komatsushima, Tokushima
  - Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - Boehringer Ingelheim Investigational Site, Koriyama,Fukushima
  - Boehringer Ingelheim Investigational Site, Kounan, Aichi
  - Boehringer Ingelheim Investigational Site, Kumagaya, Saitama
  - Boehringer Ingelheim Investigational Site, Kurashiki, Okayama
  - Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - Boehringer Ingelheim Investigational Site, Matsuyama, Ehime
  - Boehringer Ingelheim Investigational Site, Minato-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Musashino, Tokyo
  - Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - Boehringer Ingelheim Investigational Site, Nakano-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Nangoku, Kochi
  - Boehringer Ingelheim Investigational Site, Nishinomiya, Hyogo
  - Boehringer Ingelheim Investigational Site, Noda, Chiba
  - Boehringer Ingelheim Investigational Site, Nomi, Ishikawa
  - Boehringer Ingelheim Investigational Site, Obihiro, Hokkaido
  - Boehringer Ingelheim Investigational Site, Odawara, Kanagawa
  - Boehringer Ingelheim Investigational Site, Oita, Oita
  - Boehringer Ingelheim Investigational Site, Okawa, Fukuoka
  - Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - Boehringer Ingelheim Investigational Site, Osaka
  - Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - Boehringer Ingelheim Investigational Site, Osaka-sayama, Osaka
  - Boehringer Ingelheim Investigational Site, Otaru, Hokkaido
  - Boehringer Ingelheim Investigational Site, Oyama, Tochigi
  - Boehringer Ingelheim Investigational Site, Sagamihara, Kanagawa
  - Boehringer Ingelheim Investigational Site, Sakai, Osaka
  - Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - Boehringer Ingelheim Investigational Site, Setagaya-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Seto, Aichi
  - Boehringer Ingelheim Investigational Site, Shibetsu, Hokkaido
  - Boehringer Ingelheim Investigational Site, Shibuya-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Shinagawa, Tokyo
  - Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Shinjyuku-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Shiojiri, Nagano
  - Boehringer Ingelheim Investigational Site, Sunagawa, Hokkaido
  - Boehringer Ingelheim Investigational Site, Takamatsu, Kagawa
  - Boehringer Ingelheim Investigational Site, Takarazuka, Hyogo
  - Boehringer Ingelheim Investigational Site, Takasaki, Gunma
  - Boehringer Ingelheim Investigational Site, Takatsuki, Osaka
  - Boehringer Ingelheim Investigational Site, Tama, Tokyo
  - Boehringer Ingelheim Investigational Site, Toride, Ibaraki
  - Boehringer Ingelheim Investigational Site, Tosu, Saga
  - Boehringer Ingelheim Investigational Site, Toyohashi, Aichi
  - Boehringer Ingelheim Investigational Site, Toyota, Aichi
  - Boehringer Ingelheim Investigational Site, Tsuchiura, Ibaraki
  - Boehringer Ingelheim Investigational Site, Tsuchiura,Ibaraki
  - Boehringer Ingelheim Investigational Site, Tsukuba, Ibaragi
  - Boehringer Ingelheim Investigational Site, Uji, Kyoto
  - Boehringer Ingelheim Investigational Site, Ushiku, Ibaraki
  - Boehringer Ingelheim Investigational Site, Uwajima, Ehime
  - Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa